CLINICAL TRIAL: NCT05334992
Title: Reducing Pre-Death Grief, Burden, and Stress in Informal Caregivers: A Group and Individual Therapy Approach
Brief Title: Improving Mental Health for Care Partners of Persons With AD/ADRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TexasTechU; tech (Other: TexasTechU)
Record Dates: First submitted 2022-03-21; First posted 2022-04-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue; Grief; Burden, Caregiver
MeSH Terms: conditions — Caregiver Burden | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Mindfulness Based Cognitive Therapy; Behavior Activation; Group Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): Mindfulness-Based Cognitive Therapy (MBCT) combines the ideas of cognitive therapy with meditative practices and attitudes based on the cultivation of mindfulness. The heart of this work lies in becoming acquainted with the modes of mind that often characterize mood disorders while simultaneously learning to develop a new relationship to them.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Behavior Activation (Experimental): BA Increase reinforcing behaviors in order to influence emotions and cognitions.
  Interventions: Behavioral: Behavior Activation

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Individual therapy 12 to 16 weeks
  Other Names: MBCT
  Arms: Mindfulness Based Cognitive Therapy
Behavioral: Behavior Activation — Individual therapy 12 to 16 weeks
  Other Names: BA
  Arms: Behavior Activation

SUMMARY:
The overarching goal of this project is to evaluate if evidence-based interventions can reduce PDG, burden, and stress in informal caregivers of individuals with dementia

DETAILED DESCRIPTION:
Aim 1: Examine the effects of two individual evidence-based therapies for informal caregivers of dementia patients.

Aim 2: Examine the effects of a modified evidence-based group therapy for informal caregivers of dementia patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be informal caregivers (e.g., spouse; child; close friend) of individuals with dementia
* Informal caregivers can be family members or close friends
* Adults (18 to 89 years old) who read, write, and speak in English
* Mental Health Diagnosis (e.g., Generalized Anxiety Disorder; Major Depressive Disorder

Exclusion Criteria:

* Formal caregivers (who are being paid to take care of the patient)
* Any informal caregivers with cognitive impairment is identified during the assessment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief Scale-12 (measuring pre-death grief) | through study completion, an average of 6 months
  The PG-12 (range 11-55; higher scores mean higher pre-death grief), which is used to measure pre-death grief will be used to measure grief of having a loved one live with a life limiting illness and no longer be able to engage in valued activites.

SECONDARY OUTCOMES:
Zarit Burden Inventory (ZBI) | through study completion, an average of 6 months
  Informal caregivers, usually family member, have an increase in burden or feeling they are overwhelmed by their current circumstances. The ZBI is between 0-48, higher scores indicating higher burden.
Perceived Stress Scale | through study completion, an average of 6 months
  Informal caregivers, usually family members, are unpaid and have a tendency to feel tense and emotionally drained do to caregiving. Scores range from 0-40 with higher scores indicating higher rates of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Singer, Ph.D, Principal Investigator — jonsinge@ttu.edu
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No